CLINICAL TRIAL: NCT07129018
Title: A Prospective, Open-Label, Multicenter Phase II Clinical Study of Trastuzumab Rezetecan Combined With Pertuzumab and Iparomlimab and Tuvonralimab as First-Line Therapy for HER2-Expressing Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: Trastuzumab Rezetecan Combined With Pertuzumab and Iparomlimab and Tuvonralimab for Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HER2-TRIP
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer (BTC); First-line Therapy
Keywords: Iparomlimab and Tuvonralimab; Pertuzumab; Trastuzumab-rezetecan; HER2-expressing; biliarytract cancer (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HER2 Overexpression Cohort (Experimental): HER2 Overexpression ：IHC 3+ or IHC 2+/FISH +；
  Interventions: Drug: Trastuzumab-rezetecan + Pertuzumab + Iparomlimab and Tuvonralimab for HER2 Overexpression BTC
- HER2 Moderate/Low Expression Cohort (Experimental): HER2 Moderate/Low Expression：IHC 2+/FISH -（Moderate Expression）IHC 1+（Low Expression）；
  Interventions: Drug: Trastuzumab-rezetecan + Pertuzumab + Iparomlimab and Tuvonralimab for HER2 Moderate/Low BTC

INTERVENTIONS:
Drug: Trastuzumab-rezetecan + Pertuzumab + Iparomlimab and Tuvonralimab for HER2 Overexpression BTC — Subjects received treatment with Iparomlimab and Tuvonralimab (5.0 mg/kg, iv, d1, q3w) and Trastuzumab-rezetecan (4.8 mg/kg, iv, d1, q3w) in combination with Pertuzumab (initial dose 840 mg, iv, followed by 420 mg, iv, d1, q3w). Study treatment continued until the occurrence of a protocol-specified treatment discontinuation event. Following the end of treatment, subjects will continue to undergo safety follow-up and survival follow-up. For subjects who discontinued treatment for reasons other than disease progression, periodic tumor imaging assessment follow-up will also continue after treatment cessation.
  Other Names: Three-drug combination regimen
  Arms: HER2 Overexpression Cohort
Drug: Trastuzumab-rezetecan + Pertuzumab + Iparomlimab and Tuvonralimab for HER2 Moderate/Low BTC — Subjects received treatment with Iparomlimab and Tuvonralimab (5.0 mg/kg, iv, d1, q3w) and Trastuzumab-rezetecan (4.8 mg/kg, iv, d1, q3w) in combination with Pertuzumab (initial dose 840 mg, iv, followed by 420 mg, iv, d1, q3w). Study treatment continued until the occurrence of a protocol-specified treatment discontinuation event. Following the end of treatment, subjects will continue to undergo safety follow-up and survival follow-up. For subjects who discontinued treatment for reasons other than disease progression, periodic tumor imaging assessment follow-up will also continue after treatment cessation.
  Other Names: Three-drug combination regimen
  Arms: HER2 Moderate/Low Expression Cohort

SUMMARY:
Based on unmet clinical needs, relevant research backgrounds, and scientific evidence, it is planned to conduct a prospective, dual-cohort exploratory study. The aim of this study is to explore the efficacy and safety of ricartuzumab combined with pertuzumab and epalrestat-vorolizumab in the first-line treatment of HER2-expressing locally advanced or metastatic biliary tract cancer. It is expected to provide more treatment options for biliary tract cancer patients, optimize treatment strategies, and improve patients' long-term survival rates.

DETAILED DESCRIPTION:
The aim of this study is to explore the efficacy and safety of ricartuzumab combined with pertuzumab and epalrestat-vorolizumab in the first-line treatment of HER2-expressing locally advanced or metastatic biliary tract cancer. It is expected to provide more treatment options for biliary tract cancer patients, optimize treatment strategies, and improve patients' long-term survival rates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must voluntarily participate in the trial, provide fully informed consent with signed written documentation, and demonstrate good compliance.
2. Age between 18 and 75 years (inclusive), calculated as of the day of signing the informed consent form; both male and female patients are eligible.
3. Patients must have histologically or cytologically confirmed locally advanced or metastatic biliary tract cancer, including: Cholangiocarcinoma (intrahepatic or extrahepatic) and Gallbladder carcinoma
4. HER2 Expression Criteria: HER2 Overexpression: IHC 3+ OR IHC 2+ with FISH-positive (gene amplification); HER2 Moderate/Low Expression: Moderate: IHC 2+ with FISH-negative (no gene amplification) Low: IHC 1+ (any level of HER2 staining)
5. Patients must not have received prior systemic anti-tumor therapy for advanced disease. Prior neoadjuvant/adjuvant chemotherapy and/or radiotherapy is permitted, provided ≥6 months have elapsed between the last dose and disease recurrence.
6. Patients must have at least one measurable lesion meeting RECIST v1.1 criteria, and the lesion must be suitable for repeated accurate measurements.
7. ECOG performance status of 0 or 1;
8. estimated life expectancy ≥12 weeks;
9. Adequate organ and bone marrow function meeting all criteria below (within 14 days prior to treatment initiation): 1. Hematological Tests *(No transfusion, G-CSF use, or corrective medication within 14 days before screening)* Hemoglobin (Hb) ≥90 g/L Absolute Neutrophil Count (ANC) ≥1.5 × 10<sup>9</sup>/L Platelets (PLT) ≥75 × 10<sup>9</sup>/L 2. Biochemical Tests (No albumin infusion within 14 days before screening) Total Bilirubin (TBIL) ≤2 × ULN Gilbert's syndrome: ≤3 × ULN ALT/AST ≤3.0 × ULN Liver metastasis: ≤5 × ULN Serum Creatinine (Cr) ≤1.5 × ULN OR Creatinine Clearance (CrCl) ≥50 mL/min (Cockcroft-Gault formula);
10. Patients with detectable HBV DNA levels (≥10 IU/mL or above the lower limit of quantification per local laboratory assays) who are HBV-infected (HBsAg-positive and/or anti-HBc-positive) must receive antiviral therapy prior to treatment initiation according to institutional practice to achieve sufficient viral suppression. Antiviral therapy must be maintained throughout the study and for 6 months after the last dose of study treatment. Patients with positive anti-HBc but undetectable HBV DNA (<10 IU/mL or below the lower limit of quantification per local laboratory assays) do not require antiviral prophylaxis unless HBV DNA exceeds 10 IU/mL or reaches detectable levels during treatment monitoring.
11. Childbearing potential females: Negative pregnancy test (urine/serum) within 7 days pre-dose (serum result definitive if urine inconclusive). Sexually active with non-sterilized males: Use acceptable contraception from screening until 120 days post-last dose.
12. Non-sterilized males sexually active with childbearing-potential partners: Use effective contraception from screening until 120 days post-last dose. Discontinuation post-120 days requires investigator discussion.
13. Subjects must comply with visits, treatment, lab tests, and study requirements.

Exclusion Criteria:

1. Histologically or cytologically confirmed ampullary carcinoma, small cell carcinoma, neuroendocrine tumors, sarcoma, mucinous cystic neoplasms, or other rare biliary tract malignancies.
2. Active other malignancies within 5 years or concurrently.
3. History of leptomeningeal disease, brain metastases, or current brain metastases.
4. Participation in other investigational drug trials within the past 3 months, or concurrent enrollment in another interventional clinical trial (observational/non-interventional studies or follow-up phases allowed).
5. Any condition deemed by the investigator to compromise safety or compliance, including: Uncontrolled systemic diseases (e.g., severe hypertension, moderate/severe symptomatic ascites) Uncontrolled/moderate-or-greater pleural/pericardial effusion Acute/chronic uncontrolled pancreatitis Active bleeding disorders, infections, or ILD/interstitial lung disease Severe chronic GI disorders with diarrhea Psychiatric illness/social circumstances affecting compliance History of allogeneic organ or bone marrow transplantation.
6. Within 12 months prior: NYHA Class ≥II congestive heart failure Unstable angina, myocardial infarction Poorly controlled arrhythmia or cerebrovascular accident LVEF <50% by echocardiogram QTc >480 ms (Fridericia method; average of 3 measurements if abnormal) Uncontrolled hypertension (SBP≥150 mmHg and/or DBP≥100 mmHg, average of ≥2 readings) History of hypertensive crisis or encephalopathy.
7. Active autoimmune disease within 2 years or history of recurrent autoimmune disease (e.g., autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyper/hypothyroidism). (Except hypothyroidism controlled by hormone replacement)
8. Previous treatment with HER2-targeted agents, HER2-ADCs, or immunotherapy (e.g., checkpoint inhibitors/agonists, cell therapy). Therapeutic cancer vaccines excluded.
9. Prior anti-tumor therapy toxicities not recovered to CTCAE v5.0 Grade ≤1 (alopecia/lab abnormalities meeting inclusion criteria allowed per investigator).
10. Unexplained intra-abdominal gas unrelated to recent surgery/paracentesis.
11. Abdominal complications within 6 months: Abdominal fistula, gastrointestinal perforation, or abscess；Tumor invasion of adjacent organs (e.g., aorta, trachea) with high bleeding/fistula risk.
12. Immunodeficiency (e.g., HIV infection) or history of organ transplantation.
13. Active tuberculosis (TB): Active TB within 1 year prior to enrollment；Untreated active TB history >1 year prior.
14. Bleeding/thrombotic risks: Gastrointestinal bleeding within 6 months or high bleeding tendency；Known hereditary/acquired bleeding disorders or thrombophilia.
15. Surgical history: Major surgery within 4 weeks prior (excluding biopsies) or unhealed surgical wounds ；Planned major surgery during the study；Minor traumatic surgery within 7 days prior；
16. Severe/unhealed wounds, active ulcers, or untreated fractures.
17. CNS metastases (past or present).
18. Live attenuated vaccines: Administered within 28 days before the first study dose; Planned use during the study or within 60 days after the last dose.
19. Other exclusionary factors per investigator judgment (e.g., substance abuse, severe comorbidities, abnormal lab values, psychosocial circumstances).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by RECIST1.1 | Up to approximately 4 years
  Objective Response Rate (ORR) assessed by investigators based on the Response EvaluationCriteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by mRECIST | Up to approximately 4 years
  Objective Response Rate (ORR) assessed by investigators based on the modified Response Evaluation Criteria in Solid Tumors mRECIST.
DCR | Up to approximately 4 years
  The percentage of subjects who achieved complete response, partial response, or stable disease (SD) lasting for 6 weeks or longer, as determined by the investigator in accordance with RECIST v1.1 or mRECIST.
OS | Up to approximately 4 years
  The time from the date of the first drug administration to the death of the subject due to various reasons.
TTP | Up to approximately 4 years
  The time from the date of the first treatment to the occurrence of radiological disease progression, as determined by the investigator in accordance with RECIST v1.1 or mRECIST.
DoR | Up to approximately 4 years
  The time from the first documentation of objective response (CR or PR) to the first occurrence of radiological disease progression or death (whichever comes first), as determined by the investigator in accordance with RECIST v1.1 or mRECIST.
PFS | Up to approximately 4 years
  The time from the first treatment to the first occurrence of radiological disease progression or death (whichever comes first), as determined by the investigator in accordance with RECIST v1.1 or mRECIST.
Incidence of Adverse Events (AEs) | Up to approximately 4 years
  The percentage of patients in the safety analysis set who experienced specific adverse events during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Jun Xue, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Feng Shen, Principal Investigator — Eastern Hepatobiliary Surgery Hospital

IPD SHARING:
Plan to Share IPD: No